CLINICAL TRIAL: NCT05541679
Title: Comparison of Left Bundle Branch Area Versus Right Ventricular Septal Pacing in Patients With High-degree Conduction Disease After Transcatheter Aortic Valve Replacement
Brief Title: Comparison of Left Bundle Branch Area Versus Right Ventricular Septal Pacing in Patients With High-degree Conduction Disease After Transcatheter Aortic Valve Replacement (Left Bundle BRAVE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Main Line Health (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-22-5212
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Complete Heart Block; High Degree Second Degree Atrioventricular Block; Pacemaker-Induced Cardiomyopathy; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Device: Right ventricular septal pacing followed by left bundle branch area pacing
- Group B (Experimental)
  Interventions: Device: Left bundle branch area pacing followed by right ventricular septal pacing

INTERVENTIONS:
Device: Right ventricular septal pacing followed by left bundle branch area pacing — All patients will undergo implantation of right ventricular septal lead, left bundle branch area lead, and atrial lead in the absence of permanent atrial fibrillation with a CRT-pacing generator. Patients will be randomized to pacing protocols based on group assignment and crossover during the study.
  Arms: Group A
Device: Left bundle branch area pacing followed by right ventricular septal pacing — All patients will undergo implantation of right ventricular septal lead, left bundle branch area lead, and atrial lead in the absence of permanent atrial fibrillation with a CRT-pacing generator. Patients will be randomized to pacing protocols based on group assignment and crossover during the study.
  Arms: Group B

SUMMARY:
The purpose of the study is to investigate the superiority of chronic left bundle branch area pacing compared to traditional right ventricular (RV) septal pacing in patients with high-grade conduction disease after transcatheter aortic valve replacement (TAVR). In this investigator initiated, multicenter, prospective, double-blinded, crossover study, chronic left bundle branch area pacing will be compared to chronic right ventricular septal pacing using echocardiographic measures of left ventricular systolic function in patients with a high cumulative ventricular pacing burden after TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Subject has at least one of these conduction disturbances:

  1. Symptomatic (or hemodynamically significant) bradycardia or symptomatic persistent atrioventricular block including first-degree and Mobitz I (Wenckebach) or Mobitz type II atrioventricular bock
  2. High-grade atrioventricular block
  3. Third-degree atrioventricular block
* Subject has undergone TAVR (any valve system) in the last four weeks
* Subject is receiving a first-time pacemaker implant
* Subject's most recent documented ejection fraction (by any method) within the past 90 days prior to study enrollment is > 50% (≥45% if visually estimated at the time of enrollment)
* Subject is a male or female at least 18 years old at the time of consent
* Subject is able to receive a left sided pectoral implant

Exclusion Criteria:

* Subject has ever had a previous or has an existing implantable pulse generator (IPG), implantable cardiac defibrillator (ICD) or biventricular (BiV) implant
* Subject has more than mild para-valvular regurgitation following TAVR implantation.
* Subject has LVEF < 45% if visually estimated at the time of enrollment
* Subject is indicated for a biventricular pacing device (CRT-P or CRT-D).
* Subject is enrolled in a concurrent study that may confound the results of this study
* Subject has a mechanical heart valve
* Subject is pregnant, or of childbearing potential and not on a reliable form of birth control
* Subject status post heart transplant
* Subject life expectancy less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in global longitudinal strain (GLS%) | 9 months
  Primary efficacy outcome
Change in left ventricular ejection fraction (LVEF%) | 9 months
  Primary efficacy outcome
Composite of left bundle branch area pacing lead septal myocardial or coronary artery perforation, lead dislodgment, and repeat procedures related to left bundle branch area lead implantation | 18 months
  Primary safety endpoint

SECONDARY OUTCOMES:
Adverse events related to device function | 18 months
Quality of life measured using the Minnesota Living with Heart Failure questionnaire (MLHQ) | 9 months
Functional capacity measured using the New York Heart Association functional classification (NYHA) | 9 months
Six minute walk test score | 9 months
Hospitalizations for heart failure | 18 months
Mortality | 18 months
Right ventricular global longitudinal strain (RVGLS%) | 9 months
Left ventricular mechanical systolic dyssynchrony indexed to heart rate (SDI) | 9 months
Interventricular mechanical delay (IVMD) | 9 months
Left ventricular end-systolic volume | 9 months
Left ventricular stroke volume | 9 months
Severity of tricuspid regurgitation | 18 months
Severity of mitral regurgitation | 18 months
Left bundle branch area pacing lead pacing threshold | 18 months
Left bundle branch area pacing lead sensed R wave amplitude | 18 months
Left bundle branch area pacing lead impedence | 18 months
Brain natriuretic peptide or N-terminal pro-brain natriuretic peptide concentration | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keramati, MD, Principal Investigator — Lankenau Heart Institute
Locations (4):
- United States (4):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Valley Health System, Ridgewood, New Jersey
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liskov S, Olleik F, Jarrett H, Abramson S, Kowey P, Schaller RD, Vijayaraman P, Habibi M, Bansal S, Heimann M, Cox S, Keramati AR. Comparing Left Bundle Branch Area vs Right-Ventricular Septal Pacing in High-Degree Conduction Disease After Transcatheter Aortic Valve Replacement: Randomized Trial Study Protocol. CJC Open. 2024 May 18;6(9):1058-1065. doi: 10.1016/j.cjco.2024.05.006. eCollection 2024 Sep. PMID 39525828